CLINICAL TRIAL: NCT03224013
Title: Hyperopic LASIK With Concurrent Prophylactic High-fluence Cross-linking Versus Standard LASIK Outcomes
Brief Title: Hyperopic LASIK With Crosslinking Versus Standard LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahemd Abdelghany, Lecturer of Ophthalmology.Faculty of Medicine, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Hyperopic LASIK
Record Dates: First submitted 2017-07-15; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hyperopia
MeSH Terms: conditions — Hyperopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Intervention Model Description: Interventional prospective consecutive comparative case control series of cases; 50 eyes of 25 patients with mean age 35.7 ± 12.4 (Range 18-61years) with hyperopia or hyperopic astigmatism underwent customized LASIK with concurrent prophylactic high-fluence cross-linking in right eye (group 1) and customized LASIK only in left eye (group 2). Cases with hyperopia +1D to +6D or hyperopic astigmatism up to 4D were included in the study. Patients with previous intraocular or corneal surgery, active corneal disease were excluded from the study.
  Main outcome measures were uncorrected visual acuity (UCVA), manifest refractive spherical equivalent (MRSE), cycloplegic refractive spherical equivalent (CRSE), keratometric measurments and spherical aberrations at 4 mm and maximum pupilnand their ecolution along 6 months postoperatively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperopic LASIK with crosslinking (Active Comparator): group 1:hyperopic customized LASIK with concurrent prophylactic high-fluence cross-linking
  Interventions: Procedure: LASIK
- Hyperopic LASIK only (Active Comparator): group 2: hyperopic customized LASIK only
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — LASIK with concurrent prophylactic high fluence crosslinking in right eye ( After the excimer laser ablation, and with the flap folded onto itself and protected with a dry sponge, one drop of Vibex Rapid™ , consisting of 0.10% saline-diluted riboflavin (a very slightly hypotonic solution, mixed with hydroxypropyl methylcellulose, a dextran substitute), was placed on the exposed stromal bed afforded by the open LASIK flap and carefully spread over the bed area with an irrigating cannula for 60 seconds and LASIK only in left eye

SUMMARY:
Analysis corneal and refractive stability of hyperopic laser-assisted in situ keratomileusis (LASIK) with and without concurrent prophylactic high-fluence cross-linking (CXL).

DETAILED DESCRIPTION:
Interventional prospective consecutive comparative case control series of cases; 50 eyes of 25 patients with mean age 35.7 ± 12.4 (Range 18-61years) with hyperopia or hyperopic astigmatism underwent customized LASIK with concurrent prophylactic high-fluence cross-linking in right eye (group 1) and customized LASIK only in left eye (group 2). Cases with hyperopia +1 diopter to +6 diopters or hyperopic astigmatism up to 4 diopters were included in the study. Patients with previous intraocular or corneal surgery, active corneal disease were excluded from the study.

Main outcome measures were uncorrected visual acuity (UCVA), manifest refractive spherical equivalent (MRSE), cycloplegic refractive spherical equivalent (CRSE), keratometric measurements and spherical aberrations at 4 mm and maximum pupil and their evolution along 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Cases with hyperopia +1diopter to +6 diopters or hyperopic astigmatism up to 4 diopters

Exclusion Criteria:

* Patients with previous intraocular or corneal surgery, active corneal disease

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
assessment of changes in refractive spherical equivalent | preoperative and 3 months and 6 months postoperative
  assessment of changes in manifest refraction by autorefractometer and then calculate spherical equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L Alio, MD, Study Director — MD, Phd, FEBO

IPD SHARING:
Plan to Share IPD: No